CLINICAL TRIAL: NCT04242979
Title: Assessing of Physicians' Knowledge About International Guidelines of Albumin Use in Patients With Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abdelrahman Salah Eldin Abodief (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Salah Eldin Abodief, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HA use in liver cirrhosis
Record Dates: First submitted 2020-01-11; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Liver Cirrhoses
Keywords: Albumin use in liver cirrhosis

STUDY DESIGN:
Intervention Model Description: Tool (I):
  An interview questionnaire(in English) sheet for the physicians will be carried out evaluating :
  1. the use of albumin in validated indications.
  2. the prescriptions of albumin for non validated clinical situations.
  TOOL (II):
  Designed evidence-based indications for HA use supported by the international guidelines.
  It includes general information about albumin prescription, mechanism of action of albumin in liver cirrhosis, prevention of PPCD, prevention of renal failure after SBP, diagnosis of HRS, treatment of HRS, other potential clinical indication for albumin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human albumin use in liver cirrhosis (Other): Each participant involved in the study will be assessed for his or her knowledge using (tool I).
  5-Data will be collected by personal interview with participants or via fulfilling online questionnaire taking in consideration data confidentiality.
  6-Application of the designed evidence based indications for human albumin use supported by the international guidelines will be done by researcher using (tool II).
  7-Evaluate the effect of the designed evidence based indications for human albumin use supported by the international guidelines on physicians' knowledge after 1 month using (tool I) in a random sample of those physicians.
  Interventions: Behavioral: Questionnaire about albumin use in liver cirrhosis

INTERVENTIONS:
Behavioral: Questionnaire about albumin use in liver cirrhosis — 1. Permission to carry out the study will be obtained from the Faculty's Ethics Committee.
  2. To achieve validity and reliability of the tool. It will be reviewed by two experts in the field of the study and necessary modification will be done.
  3. A pilot study will be 10% done to test the clarity and feasibility of developed tool.
  4. Each participant involved in the study will be assessed for his or her knowledge using (tool I).
  5. Data will be collected by personal interview with participants or via fulfilling online questionnaire taking in consideration data confidentiality.
  6. Application of the designed evidence based indications for human albumin use supported by the international guidelines will be done by researcher using (tool II).
  7. Evaluate the effect of the designed evidence based indications for human albumin use supported by the international guidelines on physicians' knowledge after 1 month using (tool I) in a random sample of those physicians

SUMMARY:
Due to shortage of local studies of the adherence of physicians to the guidelines for albumin use among patients with liver cirrhosis so this study aims to assess:

1. Physicians' knowledge on the evidence-based indications for HA use supported by the international guidelines;
2. Whether HA is used in clinical conditions not supported by solid scientific evidence;
3. To formulate the evidence-based indications for HA use supported by the international guidelines and to evaluate effect of distributing these evidence-based indications on physicians' knowledge.

DETAILED DESCRIPTION:
* In the last part of the previous century the increasing knowledge about the cardiovascular abnormalities that occur in advanced cirrhosis led researchers to design prospective randomized clinical trials assessing the effect of exogenous human albumin (HA) based on its well-established capacity to act as plasma-expander.
* Due to the positive results reported by those studies, international guidelines have included the administration of HA among the recommendations for the prevention of post-paracentesis circulatory dysfunction (PPCD) or renal failure induced by spontaneous bacterial peritonitis (SBP), and for the diagnosis and treatment of hepatorenal syndrome (HRS) .
* Indeed, all these complications are characterized by a substantial reduction of effective volemia. However, even in these settings, questions regarding HA dosage and whether or not all patients should be treated remain unanswered .
* It has now become evident that circulatory dysfunction and organ damage in patients with decompensated cirrhosis are related to a chronic state of systemic inflammation and oxidative stress, which can abruptly exacerbate in patients developing acute-on-chronic liver failure (ACLF), a syndrome characterized by extra-hepatic organ failure and poor short-term survival.
* Besides colloid-osmotic power, HA is provided with many biological properties unrelated to the regulation of fluid compartmentalization. Among these, some would assume particular importance in relation to the inflammatory state of decompensated cirrhosis, such as antioxidant and scavenging activities, binding and transport of many endogenous and exogenous substances, and regulation of endothelial function and inflammatory/immunological response .
* Therefore, due to both its oncotic and non-oncotic properties, HA may exert beneficial effects at different steps of the cascade of the pathogenetic events that link circulatory dysfunction to systemic inflammation, providing a novel pathophysiological perspective for the use of HA. In this regard, two nationwide surveys on the use of HA in patients with cirrhosis conducted in the United States and France aiming to assess the adherence to the current AASLD and EASL guidelines respectively, have shown that HA is also prescribed besides the evidence-based indications. Indeed, HA is not rarely employed in non-SBP bacterial infections, severe hyponatremia, and hypoalbuminemia.

ELIGIBILITY:
Inclusion Criteria:

Gastroenterology physicians in:

* Al-Rajhi Liver Hospital (Tropical Medicine Department, and Internal Medicine, GIT Unit).
* Police Hospital.
* Health Insurance Hospital.
* Assiut Center for Management of HCV.
* El - Shamla Hospital.
* Al-Eman Hospital.

Exclusion Criteria:

* Non gastroenterology physicians

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | 1 month
  The investigators will know physicians' basic mean knowledge score about human albumin use in validated and non validated indications.
  The score will be from (0-2)

SECONDARY OUTCOMES:
Questionnaire | 2-3 years
  The investigators will determine the effect of designed evidence based indication for human albumin use supported by the international guidelines on mean knowledge scores of physicians.The score will be from (0-2)

REFERENCES:
- [Background] Caraceni P, Pavesi M, Baldassarre M, Bernardi M, Arroyo V. The use of human albumin in patients with cirrhosis: a European survey. Expert Rev Gastroenterol Hepatol. 2018 Jun;12(6):625-632. doi: 10.1080/17474124.2018.1460203. Epub 2018 Apr 4. PMID 29611452